CLINICAL TRIAL: NCT01793090
Title: Phase 2, Double-Blind, Placebo Controlled Clinical Trial of EPI-743 in Subjects With Cobalamin C Defect
Brief Title: EPI-743 in Cobalamin C Defect: Effects on Visual and Neurological Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giancarlo Iarossi, MD, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-12-92
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Methylmalonic Aciduria and Homocystinuria,Cblc Type; Genetic Disease; Retinopathy
Keywords: Cobalamin C defect; methylmalonic aciduria with homocystinuria; Visual function; VEP; ERG; antioxidant drugs
MeSH Terms: conditions — Methylmalonic acidemia with homocystinuria; Genetic Diseases, Inborn; Retinal Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPI-743 (Active Comparator): EPI- 743 in capsule or formulation comprised of USP/NF (United States Pharmacopeia and The National Formulary)Sesame Oil at a potency of 100 mg EPI-743/ 1 mL total volume. Mode of Administration: Oral with meal or G-Tube infusion with food.
  Dose: 100mg or 200 mg tid for 12 months, to be continued if clinically effective
  Interventions: Drug: Epi-743
- Placebo supplementation (Placebo Comparator): placebo in the same formulation as the active comparator will be administered to patients, assigned to this arm in a randomized design
  Interventions: Other: Placebo supplementation

INTERVENTIONS:
Drug: Epi-743 — EPI- 743 in capsule or formulation comprised of USP/NF Sesame Oil at a potency of 100 mg EPI-743/ 1 mL total volume. Mode of Administration: Oral with meal or G-Tube infusion with food.
  Arms: EPI-743
Other: Placebo supplementation — Placebo will be administered in the same formulation as the active comparator
  Arms: Placebo supplementation

SUMMARY:
The aim of the research is to investigate the safety and efficacy of EPI-743 treatment in patients with Cbl-C defect and related visual and neurological impairment. Primary Endpoints will be the improvement in visual function as assessed by visual acuity and eye-hand coordination and manual dexterity. Secondary Endpoints will be the improvement in neurologic function, evaluated by a battery of age-appropriated psychophysical tests, and/or in objective electrophysiological tests such as Visual Evoked potentials (VEP) and Electroretinogram (ERG) and/or the change in serum markers of redox state.

DETAILED DESCRIPTION:
Cobalamin C (Cbl-C) defect is the most common inborn error of cobalamin metabolism causing methylmalonic aciduria and homocystinuria. Cbl-Cdefect is due to impaired activity of MMACHC, a cobalamin trafficking protein, involved in the decyanation of cyanocobalamin as well as in the dealkylation of alkylcobalamins through a glutathione transferase activity. Despite pharmacological treatment with hydroxycobalamin, betaine, folic acid, (and carnitine), long-term outcome in early-onset patients is in most cases unsatisfactory with progression of visual and neurological impairment, mainly expressed in the form of retinal degeneration and/or maculopathy. Moreover, despite some hypotheses have been proposed, the pathophysiological mechanism causing progressive eye and brain damage still remains unclear. Recently, the contribution of oxidative stress has been hypothesized based on in vitro studies showing in Cbl-C fibroblasts a significant increase of reactive oxygen species (ROS) and in vivo studies documenting severe alteration of glutathione species, the main cellular redox buffer.

EPI-743 is a small molecule therapeutic that has demonstrated beneficial effects in diseases characterized by oxidative stress and alterations in glutathione redox balance including Leigh syndrome and other inherited respiratory chain diseases.

Based on the principle that Cbl-C defect causes both in vivo and in vitro perturbations of redox state, the aim of our study is to verify the potential beneficial effects of EPI-743 in preventing/reducing progression of neurological and visual signs, as well as in ameliorating redox abnormalities in Cbl-C patients, in combination with standard therapy.

Primary Endpoints will include the improvement in visual function as assessed by visual acuity and eye-hand coordination and manual dexterity. Secondary Endpoints will be improvement in neurologic function, evaluated by a battery of age-appropriated psychophysical tests, and/or in objective electrophysiological tests such as VEP and ERG, and/or the change in serum markers of redox state. Patient's and parental Quality of life will be regularly assessed prior of treatment start and periodically while on EPI-743.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed Cbl-C defect;
* abstention from antioxidant medications (i.e. coenzyme Q10, idebenone, vitamin E) prior to trial initiation and throughout conduct of trial.

Exclusion Criteria:

* allergy to EPI-743 or sesame oil (a screening test will be performed);
* abnormal coagulation;
* hepatic insufficiency with Liver Function Tests greater than 2-times normal values;
* renal insufficiency requiring dialysis;
* fat malabsorption precluding drug absorption.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Visual Function | Baseline, six months, twelve months
  Visual acuity: - Patients age 0-2: Durand acuity cards procedure: Improvement from baseline or nadir by greater than 2 lines when converted to EDTRS values.-Patients age 2-4: LEA Symbols for crowding binocular acuity: Improvement from baseline or nadir by greater than 2 lines when converted to EDTRS values; -Patients age > 4 years: Cambridge acuity cards: Improved from baseline or nadir by greater than 2 lines on the EDTRS acuity testing chart at 4 meters. Eye-hand coordination: -Patients age 0-2: Improvement over baseline of 20% on Griffiths Mental Development Scale subscales D,E; - Patients age > 2: Improvement over baseline of 20% on Movement Assessment Battery for Children

SECONDARY OUTCOMES:
Change in steady-state luminance Visual Evoked Potentials | Baseline, six months, twelve months
  Steady-state luminance VEPs to sinusoidal flicker at the optimal frequency of 8 Hz.
Evaluation of neurological function | Baseline, six months, twelve months
  Evaluation of neurological function with Gross motor function measure, movement ABC

OTHER OUTCOMES:
Biomarkers of redox state | Baseline, six months, twelve months
  Glutathione species in blood cells, Antioxidant enzymes expression, redox proteomic studies

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Dionisi-Vici, MD, Study Chair — Bambino Gesù Hospital and Research Institute; Giancarlo Iarossi, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute; Daniela Ricci, MD,PhD, Principal Investigator — Catholic University of the Sacred Heart; Diego Martinelli, MD, PhD, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy

REFERENCES:
- [Background] Martinelli D, Deodato F, Dionisi-Vici C. Cobalamin C defect: natural history, pathophysiology, and treatment. J Inherit Metab Dis. 2011 Feb;34(1):127-35. doi: 10.1007/s10545-010-9161-z. Epub 2010 Jul 15. PMID 20632110
- [Background] Nogueira C, Aiello C, Cerone R, Martins E, Caruso U, Moroni I, Rizzo C, Diogo L, Leao E, Kok F, Deodato F, Schiaffino MC, Boenzi S, Danhaive O, Barbot C, Sequeira S, Locatelli M, Santorelli FM, Uziel G, Vilarinho L, Dionisi-Vici C. Spectrum of MMACHC mutations in Italian and Portuguese patients with combined methylmalonic aciduria and homocystinuria, cblC type. Mol Genet Metab. 2008 Apr;93(4):475-80. doi: 10.1016/j.ymgme.2007.11.005. Epub 2007 Dec 27. PMID 18164228
- [Background] Ricci D, Pane M, Deodato F, Vasco G, Rando T, Caviglia S, Dionisi-Vici C, Mercuri E. Assessment of visual function in children with methylmalonic aciduria and homocystinuria. Neuropediatrics. 2005 Jun;36(3):181-5. doi: 10.1055/s-2005-865609. PMID 15944903
- [Background] Trisciuzzi MT, Riccardi R, Piccardi M, Iarossi G, Buzzonetti L, Dickmann A, Colosimo C Jr, Ruggiero A, Di Rocco C, Falsini B. A fast visual evoked potential method for functional assessment and follow-up of childhood optic gliomas. Clin Neurophysiol. 2004 Jan;115(1):217-26. doi: 10.1016/s1388-2457(03)00282-7. PMID 14706491
- [Background] Deodato F, Boenzi S, Santorelli FM, Dionisi-Vici C. Methylmalonic and propionic aciduria. Am J Med Genet C Semin Med Genet. 2006 May 15;142C(2):104-12. doi: 10.1002/ajmg.c.30090. PMID 16602092
- [Background] Carrozzo R, Dionisi-Vici C, Steuerwald U, Lucioli S, Deodato F, Di Giandomenico S, Bertini E, Franke B, Kluijtmans LA, Meschini MC, Rizzo C, Piemonte F, Rodenburg R, Santer R, Santorelli FM, van Rooij A, Vermunt-de Koning D, Morava E, Wevers RA. SUCLA2 mutations are associated with mild methylmalonic aciduria, Leigh-like encephalomyopathy, dystonia and deafness. Brain. 2007 Mar;130(Pt 3):862-74. doi: 10.1093/brain/awl389. Epub 2007 Feb 14. PMID 17301081
- [Background] Dionisi-Vici C, Deodato F, Roschinger W, Rhead W, Wilcken B. 'Classical' organic acidurias, propionic aciduria, methylmalonic aciduria and isovaleric aciduria: long-term outcome and effects of expanded newborn screening using tandem mass spectrometry. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):383-9. doi: 10.1007/s10545-006-0278-z. PMID 16763906